CLINICAL TRIAL: NCT00910364
Title: EXPERT Trial: Exercise to Prevent Post-thrombotic Syndrome Elicited by Recent Thrombosis
Brief Title: Feasibility Study of Exercise in Patients With Leg Blood Clots
Acronym: EXPERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Suman Rathbun, Professor of Medicine, University of Oklahoma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14181; ORA #20081607 (Other: Office of Research Administration)
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Deep Vein Thrombosis
Keywords: Lower extremity DVT; Clot; leg clot; Deep vein thrombosis; Thrombosis; Warfarin
MeSH Terms: conditions — Venous Thrombosis; Thrombosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise testing (Experimental): Feasibility study; all participants receive intervention
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise

SUMMARY:
The purpose of this pilot study is to assess the feasibility of determining the effects of a structured exercise program started two to four weeks after diagnosis of a first episode lower-extremity deep vein thrombosis (DVT) for a period of 12 weeks in reducing the incidence of post-thrombotic syndrome (PTS).

DETAILED DESCRIPTION:
Deep Vein Thrombosis (DVT) affects nearly 300,000 people in the U.S. each year. DVT of the leg results in PTS in up to 65% of patients,despite receiving appropriate medical management with anticoagulant therapy.

PTS, caused by persistent venous outflow obstruction and venous valvular dysfunction, may result in symptoms of leg pain, swelling, heaviness and cramping especially with prolonged standing.

All eligible patients with documented first-episode DVT interested in participating will undergo medical screening and a screening treadmill test prior to enrollment between two and four weeks post DVT diagnosis. All patients will be provided and asked to wear class II (30 to 40mmHg) knee length compression hose daily during the entire trial.

The formal exercise training includes both a supervised walking program and a home-based walking program for 12 weeks with follow-up at 26 weeks. Blood tests will be taken to measure levels of indicators of inflammation at baseline, week 4, week 12, and week 26. The primary outcomes will be the feasibility of the exercise program and the incidence of post-thrombotic syndrome at 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* First episode lower extremity DVT (proximal or distal) documented by ultrasound, CT angiogram or venogram within last 4 weeks.
* Treatment with LMWH, or unfractionated heparin (UFH) followed by warfarin adjusted to keep INR 2 to 3 for at least 3 months, or LMWH given in therapeutic doses as sole therapy.
* Age 21 to 75 years old.

Exclusion Criteria:

* Recurrent DVT.
* Treatment of DVT with systemic or catheter-directed thrombolysis Contraindications to exercise training according to the American College of Sports Medicine (e.g., acute myocardial infarction, unstable angina, etc.,).
* Life expectancy < 1 year.
* Pregnancy.
* Geographic inaccessibility.
* Screening (pre-randomization) exercise stress test demonstrating contraindication to exercise training (see exclusion #2).
* Cognitive dysfunction assessed by mini-mental status exam (score < 24).
* Inability to walk.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-10; Primary Completion 2012-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Villalta PTS score | at 26 weeks

SECONDARY OUTCOMES:
PTS, venous valvular reflux, VEINES, MOS SF-36, maximal treadmill test, 6-minute walk, and blood analysis | at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suman W. Rathbun, M.D., Principal Investigator — Oklahoma University Health Sciences Center
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States